CLINICAL TRIAL: NCT03261128
Title: Tool for the Detection of Oncogeriatric Fragility in Patients Aged ≥75 Years Undergoing Oncological Treatment. Feasibility and Acceptability Study.
Brief Title: Tool for the Detection of Oncogeriatric Fragility in Patients Aged ≥75 Years Undergoing Oncological Treatment.(D-FOG)
Acronym: D-FOG
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-A02188-45
Record Dates: First submitted 2017-08-04; First posted 2017-08-24 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: 75 Years Old and More; Cancer; Chemotherapy
Keywords: cancer; chemotherapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group D-FOG: Filling of a self-questionnaire before each chemotherapy cure
  Interventions: Other: Self-questionnaire

INTERVENTIONS:
Other: Self-questionnaire — Filling of a self-questionnaire before each chemotherapy cure

SUMMARY:
Many cancers are diagnosed after 75 years. Treatment in chemotherapy begins without evidence of geriatric risk factors. A new tool for screening for geriatric fragilities is used, a self-administered questionnaire carried out by the patient before each chemotherapy cure. The objective is to secure the quality of patient care and to detect the appearance and / or aggravation of geriatric fragilities.

DETAILED DESCRIPTION:
Evaluation of the feasibility of a new geriatric fragility screening tool (D-FOG) in patients aged ≥ 75 years during oncological treatment:

* Number of D-FOGs filled in: comparison with the number of patients included in the study and the number of visits of each patient.
* Regularity of the D-FOG self-questionnaire by the patient: comparison with the number of visits of the patient for a chemotherapy cure (HDJ or HDS).
* Number of criteria entered by D-FOG: comparison with the total number of criteria to be filled in
* Criterion analysis of D-FOG

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 75 years and over
* Carriers of diagnosed cancer (excluding hematology)
* Whatever the location, uniqueness or multiple, duration of development and treatment status (adjuvant, neoadjuvant, locally advanced or metastatic)
* Seen in nursing consultant
* Beginning an oncological treatment
* Supported for oncology day hospital (HDJ) or weekly (HDS) chemotherapy
* Patient not opposed to participate in the study

Exclusion Criteria:

* Patients under 75 years of age
* Having not had an IDE ad consultation
* During oncological treatment
* Receiving Oral Therapy or hormone therapy alone
* Treated by radiotherapy alone or surgery alone
* Not attending a day or week oncology hospital
* Refusal to participate in research

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 75 years and over Cancer and treated with chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2018-09-11 (Actual); Study Completion 2018-12-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of the feasibility of a new geriatric fragility screening tool (D-FOG) in patients aged ≥ 75 years during oncological treatment. | 3 months
  Feasibility of D-FOG for patients : number of D-FOGs filled in, regularity of the D-FOG self-questionnaire by the patient, number of criteria entered by D-FOG, criterion analysis of D-FOG

CONTACTS AND LOCATIONS:
Overall Officials: VALERO SV SIMON, Doctor, Principal Investigator — CHU Poitiers
Locations (1):
- CHU, Poitiers, France